CLINICAL TRIAL: NCT00006669
Title: Phase II Trial of EPOCH and Rituxan Combined Therapy in Patients With Refractory or Relapsed CD20 Positive Intermediate Grade B-cell Non-Hodgkin's Lymphoma
Brief Title: Rituximab Followed by Combination Chemotherapy in Treating Patients With Refractory or Recurrent Non-Hodgkin's Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068283; WHC-99365; NCI-V00-1630
Record Dates: First submitted 2000-12-06; First posted 2004-05-04 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2001-05

CONDITIONS: Lymphoma
Keywords: recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; sargramostim; EPOCH protocol; Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; Vincristine

INTERVENTIONS:
Biological: rituximab
Biological: sargramostim
Drug: EPOCH regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to kill cancer cells. Combining monoclonal antibody therapy with chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab followed by combination chemotherapy in treating patients who have refractory or recurrent non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate in patients with refractory or recurrent CD20+ intermediate grade B-cell non-Hodgkin's lymphoma treated with rituximab followed by etoposide, vincristine, doxorubicin, cyclophosphamide, and prednisone (EPOCH). II. Determine the toxicity of the regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive rituximab IV over 4-10 hours on day 1 followed by etoposide, vincristine, and doxorubicin IV continuously on days 4-7, cyclophosphamide IV over 5-30 minutes on day 8 and oral prednisone on days 4-8. Patients also receive sargramostim (GM-CSF) subcutaneously beginning on day 9 until blood counts recover. Treatment repeats every 21 days for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of intermediate grade B-cell CD20+ non-Hodgkin's lymphoma Failed to achieve initial complete response (CR) after at least 2 courses of standard chemotherapy OR Relapsed after CR and not eligible for autologous bone marrow transplant Measurable disease defined as one of the following: Bidimensionally measurable disease at least 2 cm in diameter by radiograph or CT scan Enlarged spleen extending at least 2 cm below the costal due to lymphomatous involvement Enlarged liver with focal lesions on CT scan or biopsy proven lesions Lymphomatous hepatic involvement must be biopsy proven for the liver to be sole area of measurable disease No evidence of CNS involvement A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3* Platelet count at least 100,000/mm3* *unless there is bone marrow involvement with lymphoma Hepatic: Bilirubin less than 3 mg/dL AST/ALT less than 2 times normal Renal: Creatinine less than 2.1 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: LVEF greater than 45% by MUGA or echocardiogram Other: No prior malignancy within the past 10 years except squamous cell carcinoma or basal cell carcinoma of the skin or cervical cancer No evidence of infection HIV negative Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: See Disease Characteristics No prior rituximab

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-09; Primary Completion 2000-01; Study Completion 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: Sein Aung, MD, Study Chair — Harry & Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center
Locations (2):
- United States (2):
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Franklin Square Hospital Center, Baltimore, Maryland